CLINICAL TRIAL: NCT06305481
Title: Glaucoma Evaluation With the P200TE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Optos, PLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OPT1099
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Imaging Device (Other): Various scans will be captured
  Interventions: Device: P200TE

INTERVENTIONS:
Device: P200TE — SLO and OCT imaging
  Other Names: OCT Device

SUMMARY:
Images captured on the P200TE device on glaucoma patients

ELIGIBILITY:
Inclusion Criteria

* Subjects were 22 years of age or older on the date of informed consent;
* Subjects were able to understand the written informed consent and willing to participate as evidenced by signing the informed consent;
* BCVA 20/40 or better in the study eye;
* History of visual field defects within the previous year from the study visit or measured the day of the study visit consistent with glaucomatous optic nerve damage with at least one of the following two findings:

On pattern deviation (PD), there existed a cluster of 3 or more points in an expected location of the visual field depressed below the 5% level, at least 1 of which is depressed below the 1% level; or Glaucoma hemi-field test "outside normal limits;"

-Glaucomatous optic nerve damage as evidenced by any of the following optic disc or retinal nerve fiber layer structural abnormalities: Diffuse thinning, focal narrowing, or notching of the neuroretinal rim, especially at the inferior or superior poles with or without disc hemorrhage; and Optic disc neural rim asymmetry of the two eyes consistent with loss of neural tissue.

Exclusion Criteria

* Subjects unable to tolerate ophthalmic imaging;
* Subjects with ocular media not sufficiently clear to obtain acceptable OCT images in the study eye;
* Subject has a condition or is in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study;
* No reliable visual field test result within the past year of the study visit, defined as fixation losses > 33% or false positives >33%, or false negatives >33% in the study eye;
* Presence of any ocular pathology except glaucoma in the study eye.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of images collected | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Werner Optometry, Cajon, California
  - Specialty Eyecare Centre, Bellevue, Washington